CLINICAL TRIAL: NCT04803669
Title: The Investigation of Instrument-assisted Soft Tissue Mobilization Technique on Pain and Disability in Patients With Cervical Neck Pain
Brief Title: The Effect of Instrument-assisted Soft Tissue Mobilization Technique on Neck Pain
Acronym: IASTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emresenocak (Other)
Responsible Party: Sponsor-Investigator, Emresenocak, Research Assistant, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2019.491
Record Dates: First submitted 2021-03-14; First posted 2021-03-18 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Neck Pain
Keywords: neck pain; neck disability; Instrument-assisted soft tissue mobilization technique; conventional therapy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Conventional Treatment Conventional Treatment + Instrument-assisted soft tissue mobilization technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment Group (Active Comparator): Includes Hotpack, TENS, Ultrasound and Exercise programs.
  Interventions: Procedure: Conventional Treatment
- IASTM Group (Experimental): Inludes Hotpack, TENS, Ultrasound, Exercise program and Instrument-assisted Soft Tissue Mobilization Technique
  Interventions: Procedure: Intrument-assisted soft tissue mobilization technique; Procedure: Conventional Treatment

INTERVENTIONS:
Procedure: Intrument-assisted soft tissue mobilization technique — This technique; It is applied with the help of a tool made of stainless steel. The instrument is rubbed on the skin at an angle of about 30 degrees, creating a massage-like effect on the soft tissue (2 sessions per week and 5 minutes per session, 8 sessions in total for 4 weeks).
  Arms: IASTM Group
Procedure: Conventional Treatment — Hotpack, TENS, Ultrasound and Exercise will be applied as conventional treatment methods.

SUMMARY:
In the literature, studies reporting that symptoms such as limitation of motion in the neck, reduced functionality, and disability and depression occur in cervical pain are frequently encountered. Treatments such as medical therapy, intramuscular injections, and traditional physical therapy modalities have been used in the treatment of these symptoms. In recent years, the popularity of the instrument-assisted soft tissue mobilization (IASTM) technique in the treatment of soft tissue-related problems has increased and has been widely used in studies. This technique is a low-cost, easy-to-apply, and accessible method that is frequently used in extremity soft tissue problems and trigger point treatment. The investigators did not find any study on the effectiveness of the IASTM technique on pain and functionality in cervical region disorders. For this reason, the primary purpose of the study is; While the effectiveness of the IASTM technique on pain and functionality in patients with neck pain caused by cervical disc herniation, the secondary purpose is to reveal the effect of IASTM on anxiety-depression.

DETAILED DESCRIPTION:
Ethics Approval: The study started with the approval of the Ethics Committee of Marmara University Faculty of Medicine with the 09.2019.491 protocol number.

Twenty-four patients who were diagnosed with cervical disc herniation (bulging, protrusion) based on radiological evaluation and who achieved 100% continuity in the treatment program will be included in the study. A similar study was taken as a reference when calculating the sample size.

Randomization: Participants will be randomized and divided into two groups using online randomization software. Conventional treatment methods will be applied to "Conventional Treatment Group", and IASTM will be applied to "IASTM Group" participants in addition to the conventional treatment protocol. Conventional treatment will be applied to both groups for 4 weeks, 5 days a week.

Interventions: Conventional treatment protocol was determined as hot pack application, electrotherapy agents, and exercise program. Hotpack intervention will be made on the neck and upper back area by wrapping in hot water bags and a towel for 25 minutes. The electrotherapy program consists of transcutaneous electrical stimulation (TENS) and ultrasound (US). Conventional TENS; 2 channels and 4 electrodes on the neck and upper trapezius muscle; It will be applied for 25 minutes (Acutens Brand, frequency 100 Hz, wave width 200 ms, 1-100 mA current). The current intensity will be adjusted in a way that does not cause discomfort for the patient. US will be applied at an intensity of 1-2.5 W / cm2 and a frequency of 1 MHz for 5 minutes to increase circulation in deep tissues. After the electrotherapy application, the patients will be given an exercise program under the supervision of a physiotherapist for 25 minutes. This program consists of deep flexor and extensor strengthening, posture, stretching, and mobilization exercises with elastic bands. The instrument-assisted soft tissue mobilization technique will be applied over the superficial and deep fascia region between C1-T1 neck-shoulder segments. The instrument used is made of stainless steel and will be applied using a brushing technique parallel to the muscle fibers (applications at an angle of 30 °). A water-based gel will be used to prevent adverse effects on the tissue due to friction. This technique will be applied as 2 sessions per week and 5 minutes per session, 8 sessions in total for 4 weeks.

Assessment:

* Sociodemographic Data Form: Patients' gender, age, body mass index, and time of pain onset will be noted.
* Visual Analogue Scale: The Visual Analogue Scale (VAS) is an easy-to-apply and reliable assessment scale used to determine the pain level of patients. VAS was created to digitize values that are not expressed numerically. Scoring is made between 0-10 points. "0" represents the absence of pain, "10" represents the presence of unbearable pain. Using VAS, participants will be questioned for additional information such as the time of onset of neck pain, its frequency, rest, and activity pain.
* Copenhagen Neck Functional Disability Scale: It is a valid and reliable scale that evaluates the disability of patients due to neck pain. The scale consists of 15 items. The items are answered as "Yes, No, Sometimes" and scored between 0-2 points. The total score is between 0 and 30 points. If the total score is "0", it means "no neck pain and disability", "30" means "maximum neck pain and disability".
* Hospital Anxiety and Depression Scale: It includes anxiety and depression subscales. The scale consists of 14 items in total. Even-numbered items evaluate depression, and odd-numbered items assess anxiety. Answers are in four-point Likert format and are scored between 0 and 3. The cut-off point for the anxiety subscale of the scale was reported to be 10 and 7 for the depression subscale.

Statistical Analysis: The data obtained in the study will be evaluated with SPSS 11.0 statistical program at an 80% confidence interval and p <0.05 significance level. The normal distribution of the data will be examined with the Kolmogorov Smirnov test and histogram curves.

ELIGIBILITY:
Inclusion Criteria:

* Having bulging or protruding cervical disc herniation,
* Pain severity> 2 according to VAS,
* Having neck pain complaint for at least three months

Exclusion Criteria:

* Having any neck-shoulder area injury or surgery,
* Using cortisone medication,
* Having extrusion and sequestered disc herniation,
* Being diagnosed with fibromyalgia,
* Having malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Neck Pain Changing | Change from Baseline Neck Pain at 6. week
  Pain will be evaluated with Visual Analog Scale. The scale is scored between 0 and 10. "0" means no pain, "10" means very severe pain.

SECONDARY OUTCOMES:
Neck Disability Changing | Change from Baseline Neck Disability at 6. week
  Disability will be assessed by the Copenhagen Neck Functional Disability Scale. The scale is scored between 0-30. "0" means no disability, "30" means maximum neck pain and disability.
Anxiety Changing | Change from Baseline Anxiety at 6. week
  Anxiety will be evaluated with the Hospital Anxiety and Depression Scale. High score means high anxiety.
Depression Changing | Change from Baseline Depression at 6. week
  Depression will be evaluated with the Hospital Anxiety and Depression Scale. High score means high depression.

CONTACTS AND LOCATIONS:
Overall Officials: Adem Aktürk, Medical Doktor (specialist), Principal Investigator — İstanbul Gelişim University; Mehmet Özkeskin, PhD, Principal Investigator — Ege University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No